CLINICAL TRIAL: NCT01080794
Title: Repetitive Transcranial Magnetic Stimulation (rTMS) for Motor and Mood Symptoms of Parkinson's Disease (MASTER-PD), a Multicenter Clinical Trial
Brief Title: rTMS for Motor and Mood Symptoms of Parkinson's Disease
Acronym: MASTER-PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: University of California, Los Angeles (Other); University of Florida (Other); University Health Network, Toronto (Other); The Cleveland Clinic (Other); Michael J. Fox Foundation for Parkinson's Research (Other)
Responsible Party: Principal Investigator, Alvaro Pascual-Leone, Professor of Neurology, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2010P000002
Record Dates: First submitted 2010-03-03; First posted 2010-03-04 (Estimated); Results first posted 2017-04-13 (Actual); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Parkinson's Disease; Depression
Keywords: Parkinson's Disease; Depression; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Parkinson Disease; Depression | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Double rTMS (Active Comparator): High frequency rTMS stimulation of the bilateral primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- M1 Active rTMS + DLPFC Sham rTMS (Active Comparator): High frequency stimulation of the primary motor cortex (M1) and sham stimulation of the dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- DLPFC Active rTMS + M1 Sham rTMS (Active Comparator): High frequency stimulation of the dorsolateral prefrontal cortex (DLPFC) and sham stimulation of the primary motor cortex (M1).
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)
- Double Sham rTMS (Sham Comparator): Sham rTMS stimulation of the bilateral primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC).
  Interventions: Device: Repetitive transcranial magnetic stimulation (rTMS)

INTERVENTIONS:
Device: Repetitive transcranial magnetic stimulation (rTMS) — DLPFC Active rTMS: Each treatment will consist of 2000 stimuli (50 X 4-second trains of 40 stimuli at 10 Hz, administered every 30 seconds for 25 minutes). Stimulus intensity for the first and second trains will be 80 and 90 percent of motor evoked potential (MEP), respectively. If no adverse effects are observed following each of the first two trains, then the subsequent trains will be given at MEP threshold.
  M1 Active rTMS: Stimulation will be applied one side at a time, to the motor cortex site at 90 percent of each subject's motor threshold intensity, and at a frequency of 10 Hz with 1000 stimuli per side (25 X 8-second trains of 40 stimuli).
  Sham rTMS: Patients from all four centers randomized to receive sham treatment will undergo the same procedures used in patients receiving active rTMS.
  Other Names: Transcranial Magnetic Stimulation; Noninvasive Brain Stimulation; Magstim Corporation

SUMMARY:
The purpose of this study is to determine if repetitive transcranial magnetic stimulation (rTMS), a method of noninvasive brain stimulation) is effective in the treatment of the motor (movement) and mood symptoms due to Parkinson's disease (PD).

DETAILED DESCRIPTION:
Repetitive Transcranial Magnetic Stimulation (rTMS) is a non-invasive means of brain stimulation which can produce changes to brain excitability. Following a series of daily rTMS sessions, this modulation of neural circuits and other distant effects may help some of the motor and neuropsychiatric symptoms of PD for months at a time. Recently, the FDA approved daily rTMS over the prefrontal cortex as a treatment for medication-refractory depression after demonstration of efficacy in sham-controlled trials and its safety profile. Among several small and pilot studies of rTMS in PD patients, rTMS over either the motor cortex or prefrontal cortex has been reported to show beneficial effects on motor and mood (depression) symptoms with no serious adverse events. However, the relative effectiveness of rTMS over motor, prefrontal, or both regions on both mood and motor symptoms, has yet to be established in PD patients.

We propose to conduct a four-center, blinded, sham-controlled, randomized, parallel-group study of fixed-dose, high-frequency rTMS in 160 PD patients who are experiencing depressive symptoms despite an adequate trial of at least one antidepressant. Subjects will be randomized to receive rTMS over either motor cortex, prefrontal cortex, both, or neither (sham-rTMS). Subjects will receive rTMS for 25 minutes over either the prefrontal cortex (the brain region associated with mood and depression), and/or primary motor cortex (associated with motor control), and/or sham-rTMS. After 10 days of rTMS (or sham) treatment over a 2-week period, all subjects will undergo a comprehensive assessment of motor, mood, cognition and quality of life on the first working day after the last rTMS treatment, and after 1, 3 and 6 months post-treatment. This study directly addresses the expansion of rTMS as an alternative treatment for depression in the PD population and will provide evidence as to whether motor cortex stimulation will provide additional and/or separate benefit to motor symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PD according to the UK Brain Bank Criteria, confirmed by a neurologist with expertise in movement disorders.
* Minimum of 3 years since the formal diagnosis of PD, and requiring dopaminergic therapy (at a minimum, on levodopa and/or dopamine agonist therapy).
* Minimum baseline OFF score on the motor UPDRS of 15 points of more.
* Lack of features suggestive of atypical parkinsonism, such as early prominent cerebellar, pyramidal, or autonomic dysfunction; supranuclear gaze palsy; falls within the first year of symptoms; hallucinations prior to initiating a dopaminergic agent.
* No history of neuroleptics or other drugs that induce parkinsonism in the past 60 days.
* Currently optimally treated with medications and, in the view of the treating neurologist, will unlikely be requiring anti-PD medication adjustments in the next 6 months.
* On a stable dose of all medications for 30 days (except anti-depressants- which should be stable for at least 90 days).
* Lack of dementia such that, in the view of the enrolling investigator, the patient is able to give proper informed consent. In addition, all patients must score at least a 26 out of 30 on the screening MMSE.
* HAM-D score > 12 on the first 17 questions of the scale, despite the current use of antidepressant(s) for at least 90 days, or documentation of adequate trial of antidepressants (i.e. at least 6 weeks on an optimal dose), or documentation of intolerability to antidepressants.
* Untreated depression or on a stable dose of antidepressants for 90 days (untreated patients need to have tried at least one antidepressant in the past).
* Age 21 years or older.
* Patient meets the criteria for a depressive disorder based on either the MINI interview (major depression) or SCID (minor depression, or dysthymia).

Exclusion Criteria:

* Intracranial metallic bodies (e.g. from prior neurosurgical procedure).
* Signs or symptoms of increased intracranial pressure.
* Implanted pacemaker, medication pump, vagal stimulator, deep brain stimulator, TENS unit or ventriculoperitoneal shunt.
* History of seizures or unexplained loss of consciousness.
* Possible pregnancy.
* Family history of medication refractory epilepsy.
* History of substance abuse within the last 6 months.
* History of known structural brain abnormality.
* History of exposure to repetitive TMS in the past (to minimizing risk of unblinding sham condition).
* History of exposure to ECT in the past.
* Patients with suicidal ideation deemed by the investigator to be significant enough to render the individual a suicidal risk.
* Patients with a history of hospitalization for suicidal ideation/attempts.
* Patients requiring hospitalization for their depression within the past six months will not be allowed in the study. If a participating subject's depression worsens during the study to a degree that hospitalization is deemed necessary, or if the subject develops significant suicidal ideation, he/she will be withdrawn from the study and referred to a psychiatrist for treatment.
* Patients with bipolar affective disorder and those whose depression is characterized by psychotic features.
* Patients with a history of spontaneous hallucinations or delusions as well as those with other underlying psychotic disorders (e.g., schizophrenia, schizoaffective disorder, delusional disorder). The presence of visual illusions or hallucinations deemed by the enrolling physician to be clearly related to antiparkinsonian medications will be allowed but only if the enrolling physician believes that they are stable and unlikely to require changes in medication (i.e., addition of an antipsychotic or reduction in antiparkinsonian drug dosage). Patients with delusions will be excluded.
* Subjects judged by the clinician investigator to have dementia (by DSM-IV and MMSE criteria) will be excluded.
* Subjects judged by the clinician investigator to have dementia (by MoCA criteria) will be excluded.
* Subjects with unstable medical condition such as diabetes, cardiac disease, and hypertension.
* Subjects with brittle or severe motor fluctuation that will cause severe discomfort during OFF medication testing at Baseline, immediately post-TMS, and at Months 1, 3, and 6.
* Excessive alcohol use or taking one of the following exclusionary medications: Imipramine, Amitriptyline, Doxepin, Nortriptyline, Maprotiline, Chlorpromazine, Clozapine, Foscarnet, Ganciclovir, Ritonavir, Amphetamines (MDMA, ecstasy), cocaine, phencyclidine (PCP, angel's dust), ketamine, gamma-hydroxybutyrate (GHB), theophylline, and haloperidol.

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-05; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alvaro Pascual-Leone, M.D., Ph.D., Principal Investigator — Beth Israel Deaconess Medical Center; Allan Wu, M.D., Principal Investigator — University of California, Los Angeles; Hubert Fernandez, M.D., Principal Investigator — The Cleveland Clinic; Robert Chen, BChir, MA, MB, MSc, Principal Investigator — University Health Network, Toronto; Aparna Wagle-Shukla, MD, Principal Investigator — University of Florida; Jau-Shin Lou, MD, PhD, Principal Investigator — Oregon Health and Science University
Locations (6):
- United States (5):
  - University of California Los Angeles, Los Angeles, California
  - University of Florida, Gainesville, Florida
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - The Cleveland Clinic, Cleveland, Ohio
  - Oregon Health and Science University, Portland, Oregon
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adler CH. Nonmotor complications in Parkinson's disease. Mov Disord. 2005;20 Suppl 11:S23-9. doi: 10.1002/mds.20460. PMID 15822106
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Benabid AL, Chabardes S, Seigneuret E. Deep-brain stimulation in Parkinson's disease: long-term efficacy and safety - What happened this year? Curr Opin Neurol. 2005 Dec;18(6):623-30. doi: 10.1097/01.wco.0000186839.53807.93. PMID 16280671
- [Background] Bornke Ch, Schulte T, Przuntek H, Muller T. Clinical effects of repetitive transcranial magnetic stimulation versus acute levodopa challenge in Parkinson's disease. J Neural Transm Suppl. 2004;(68):61-7. doi: 10.1007/978-3-7091-0579-5_7. PMID 15354390
- [Background] Brusa L, Versace V, Koch G, Iani C, Stanzione P, Bernardi G, Centonze D. Low frequency rTMS of the SMA transiently ameliorates peak-dose LID in Parkinson's disease. Clin Neurophysiol. 2006 Sep;117(9):1917-21. doi: 10.1016/j.clinph.2006.03.033. Epub 2006 Aug 1. PMID 16887383
- [Background] Buhmann C, Gorsler A, Baumer T, Hidding U, Demiralay C, Hinkelmann K, Weiller C, Siebner HR, Munchau A. Abnormal excitability of premotor-motor connections in de novo Parkinson's disease. Brain. 2004 Dec;127(Pt 12):2732-46. doi: 10.1093/brain/awh321. Epub 2004 Oct 27. PMID 15509619
- [Background] Burn DJ, Troster AI. Neuropsychiatric complications of medical and surgical therapies for Parkinson's disease. J Geriatr Psychiatry Neurol. 2004 Sep;17(3):172-80. doi: 10.1177/0891988704267466. PMID 15312281
- [Background] Burt T, Lisanby SH, Sackeim HA. Neuropsychiatric applications of transcranial magnetic stimulation: a meta analysis. Int J Neuropsychopharmacol. 2002 Mar;5(1):73-103. doi: 10.1017/S1461145702002791. PMID 12057034
- [Background] Cantello R. Applications of transcranial magnetic stimulation in movement disorders. J Clin Neurophysiol. 2002 Aug;19(4):272-93. doi: 10.1097/00004691-200208000-00003. PMID 12436085
- [Background] Cardoso EF, Fregni F, Martins Maia F, Boggio PS, Luis Myczkowski M, Coracini K, Lopes Vieira A, Melo LM, Sato JR, Antonio Marcolin M, Rigonatti SP, Cruz AC Jr, Reis Barbosa E, Amaro E Jr. rTMS treatment for depression in Parkinson's disease increases BOLD responses in the left prefrontal cortex. Int J Neuropsychopharmacol. 2008 Mar;11(2):173-83. doi: 10.1017/S1461145707007961. Epub 2007 Aug 21. PMID 17708780
- [Background] Chaudhuri KR, Healy DG, Schapira AH; National Institute for Clinical Excellence. Non-motor symptoms of Parkinson's disease: diagnosis and management. Lancet Neurol. 2006 Mar;5(3):235-45. doi: 10.1016/S1474-4422(06)70373-8. PMID 16488379
- [Background] Conca A, Koppi S, Konig P, Swoboda E, Krecke N. Transcranial magnetic stimulation: a novel antidepressive strategy? Neuropsychobiology. 1996;34(4):204-7. doi: 10.1159/000119312. PMID 9121622
- [Background] Crow TJ, Johnstone EC. Controlled trials of electroconvulsive therapy. Ann N Y Acad Sci. 1986;462:12-29. doi: 10.1111/j.1749-6632.1986.tb51235.x. No abstract available. PMID 2871792
- [Background] Aarsland D, Cummings JL. Depression in Parkinson's disease. Acta Psychiatr Scand. 2002 Sep;106(3):161-2. doi: 10.1034/j.1600-0447.2002.2e009.x. No abstract available. PMID 12197850
- [Background] del Olmo MF, Bello O, Cudeiro J. Transcranial magnetic stimulation over dorsolateral prefrontal cortex in Parkinson's disease. Clin Neurophysiol. 2007 Jan;118(1):131-9. doi: 10.1016/j.clinph.2006.09.002. Epub 2006 Nov 9. PMID 17097342
- [Background] Dias AE, Barbosa ER, Coracini K, Maia F, Marcolin MA, Fregni F. Effects of repetitive transcranial magnetic stimulation on voice and speech in Parkinson's disease. Acta Neurol Scand. 2006 Feb;113(2):92-9. doi: 10.1111/j.1600-0404.2005.00558.x. PMID 16411969
- [Background] Dragasevic N, Potrebic A, Damjanovic A, Stefanova E, Kostic VS. Therapeutic efficacy of bilateral prefrontal slow repetitive transcranial magnetic stimulation in depressed patients with Parkinson's disease: an open study. Mov Disord. 2002 May;17(3):528-32. doi: 10.1002/mds.10109. PMID 12112202
- [Background] Elahi B, Elahi B, Chen R. Effect of transcranial magnetic stimulation on Parkinson motor function--systematic review of controlled clinical trials. Mov Disord. 2009 Feb 15;24(3):357-63. doi: 10.1002/mds.22364. PMID 18972549
- [Background] Epstein CM. Transcranial magnetic stimulation: language function. J Clin Neurophysiol. 1998 Jul;15(4):325-32. doi: 10.1097/00004691-199807000-00004. PMID 9736466
- [Background] Epstein CM, Evatt ML, Funk A, Girard-Siqueira L, Lupei N, Slaughter L, Athar S, Green J, McDonald W, DeLong MR. An open study of repetitive transcranial magnetic stimulation in treatment-resistant depression with Parkinson's disease. Clin Neurophysiol. 2007 Oct;118(10):2189-94. doi: 10.1016/j.clinph.2007.07.010. Epub 2007 Aug 21. PMID 17714987
- [Background] Fahn S, Cohen G. The oxidant stress hypothesis in Parkinson's disease: evidence supporting it. Ann Neurol. 1992 Dec;32(6):804-12. doi: 10.1002/ana.410320616. PMID 1471873
- [Background] Fernandez HH, See RH, Gary MF, Bowers D, Rodriguez RL, Jacobson C 4th, Okun MS. Depressive symptoms in Parkinson disease correlate with impaired global and specific cognitive performance. J Geriatr Psychiatry Neurol. 2009 Dec;22(4):223-7. doi: 10.1177/0891988709335792. Epub 2009 May 8. PMID 19429848
- [Background] Fernandez HH, Tabamo RE, David RR, Friedman JH. Predictors of depressive symptoms among spouse caregivers in Parkinson's disease. Mov Disord. 2001 Nov;16(6):1123-5. doi: 10.1002/mds.1196. PMID 11748746
- [Background] Figiel GS, Epstein C, McDonald WM, Amazon-Leece J, Figiel L, Saldivia A, Glover S. The use of rapid-rate transcranial magnetic stimulation (rTMS) in refractory depressed patients. J Neuropsychiatry Clin Neurosci. 1998 Winter;10(1):20-5. doi: 10.1176/jnp.10.1.20. PMID 9547462
- [Background] Flint AJ. Epidemiology and comorbidity of anxiety disorders in the elderly. Am J Psychiatry. 1994 May;151(5):640-9. doi: 10.1176/ajp.151.5.640. PMID 8166303
- [Background] Fregni F, Santos CM, Myczkowski ML, Rigolino R, Gallucci-Neto J, Barbosa ER, Valente KD, Pascual-Leone A, Marcolin MA. Repetitive transcranial magnetic stimulation is as effective as fluoxetine in the treatment of depression in patients with Parkinson's disease. J Neurol Neurosurg Psychiatry. 2004 Aug;75(8):1171-4. doi: 10.1136/jnnp.2003.027060. PMID 15258224
- [Background] Fregni F, Simon DK, Wu A, Pascual-Leone A. Non-invasive brain stimulation for Parkinson's disease: a systematic review and meta-analysis of the literature. J Neurol Neurosurg Psychiatry. 2005 Dec;76(12):1614-23. doi: 10.1136/jnnp.2005.069849. PMID 16291882
- [Background] Friedman JH, Fernandez HH. The nonmotor problems of Parkinson's Disease. The Neurologist 6(1): 18-27, 2000.
- [Background] George MS, Wassermann EM, Kimbrell TA, Little JT, Williams WE, Danielson AL, Greenberg BD, Hallett M, Post RM. Mood improvement following daily left prefrontal repetitive transcranial magnetic stimulation in patients with depression: a placebo-controlled crossover trial. Am J Psychiatry. 1997 Dec;154(12):1752-6. doi: 10.1176/ajp.154.12.1752. PMID 9396958
- [Background] George MS, Wassermann EM, Williams WA, Callahan A, Ketter TA, Basser P, Hallett M, Post RM. Daily repetitive transcranial magnetic stimulation (rTMS) improves mood in depression. Neuroreport. 1995 Oct 2;6(14):1853-6. doi: 10.1097/00001756-199510020-00008. PMID 8547583
- [Background] Gershon AA, Dannon PN, Grunhaus L. Transcranial magnetic stimulation in the treatment of depression. Am J Psychiatry. 2003 May;160(5):835-45. doi: 10.1176/appi.ajp.160.5.835. PMID 12727683
- [Background] Ghabra MB, Hallett M, Wassermann EM. Simultaneous repetitive transcranial magnetic stimulation does not speed fine movement in PD. Neurology. 1999 Mar 10;52(4):768-70. doi: 10.1212/wnl.52.4.768. PMID 10078725
- [Background] Gill DJ, Freshman A, Blender JA, Ravina B. The Montreal cognitive assessment as a screening tool for cognitive impairment in Parkinson's disease. Mov Disord. 2008 May 15;23(7):1043-1046. doi: 10.1002/mds.22017. PMID 18381646
- [Background] Grafton ST. Contributions of functional imaging to understanding parkinsonian symptoms. Curr Opin Neurobiol. 2004 Dec;14(6):715-9. doi: 10.1016/j.conb.2004.10.010. PMID 15582373
- [Background] Ikeguchi M, Touge T, Nishiyama Y, Takeuchi H, Kuriyama S, Ohkawa M. Effects of successive repetitive transcranial magnetic stimulation on motor performances and brain perfusion in idiopathic Parkinson's disease. J Neurol Sci. 2003 May 15;209(1-2):41-6. doi: 10.1016/s0022-510x(02)00459-8. PMID 12686400
- [Background] Khedr EM, Farweez HM, Islam H. Therapeutic effect of repetitive transcranial magnetic stimulation on motor function in Parkinson's disease patients. Eur J Neurol. 2003 Sep;10(5):567-72. doi: 10.1046/j.1468-1331.2003.00649.x. PMID 12940840
- [Background] Khedr EM, Rothwell JC, Ahmed MA, Shawky OA, Farouk M. Modulation of motor cortical excitability following rapid-rate transcranial magnetic stimulation. Clin Neurophysiol. 2007 Jan;118(1):140-5. doi: 10.1016/j.clinph.2006.09.006. Epub 2006 Nov 9. PMID 17097343
- [Background] Kirsch-Darrow L, Fernandez HH, Marsiske M, Okun MS, Bowers D. Dissociating apathy and depression in Parkinson disease. Neurology. 2006 Jul 11;67(1):33-8. doi: 10.1212/01.wnl.0000230572.07791.22. PMID 16832074
- [Background] Kostic VS, Filipovic SR, Lecic D, Momcilovic D, Sokic D, Sternic N. Effect of age at onset on frequency of depression in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1994 Oct;57(10):1265-7. doi: 10.1136/jnnp.57.10.1265. PMID 7931395
- [Background] Krings T, Buchbinder BR, Butler WE, Chiappa KH, Jiang HJ, Cosgrove GR, Rosen BR. Functional magnetic resonance imaging and transcranial magnetic stimulation: complementary approaches in the evaluation of cortical motor function. Neurology. 1997 May;48(5):1406-16. doi: 10.1212/wnl.48.5.1406. PMID 9153482
- [Background] Lang AE, Obeso JA. Challenges in Parkinson's disease: restoration of the nigrostriatal dopamine system is not enough. Lancet Neurol. 2004 May;3(5):309-16. doi: 10.1016/S1474-4422(04)00740-9. PMID 15099546
- [Background] Leentjens AF. Depression in Parkinson's disease: conceptual issues and clinical challenges. J Geriatr Psychiatry Neurol. 2004 Sep;17(3):120-6. doi: 10.1177/0891988704267456. PMID 15312275
- [Background] Leentjens AF, Scholtissen B, Vreeling FW, Verhey FR. The serotonergic hypothesis for depression in Parkinson's disease: an experimental approach. Neuropsychopharmacology. 2006 May;31(5):1009-15. doi: 10.1038/sj.npp.1300914. PMID 16205779
- [Background] Lefaucheur JP, Drouot X, Von Raison F, Menard-Lefaucheur I, Cesaro P, Nguyen JP. Improvement of motor performance and modulation of cortical excitability by repetitive transcranial magnetic stimulation of the motor cortex in Parkinson's disease. Clin Neurophysiol. 2004 Nov;115(11):2530-41. doi: 10.1016/j.clinph.2004.05.025. PMID 15465443
- [Background] Lemke MR, Fuchs G, Gemende I, Herting B, Oehlwein C, Reichmann H, Rieke J, Volkmann J. Depression and Parkinson's disease. J Neurol. 2004 Sep;251 Suppl 6:VI/24-7. doi: 10.1007/s00415-004-1606-6. PMID 15675721
- [Background] Levin BE, Llabre MM, Weiner WJ. Parkinson's disease and depression: psychometric properties of the Beck Depression Inventory. J Neurol Neurosurg Psychiatry. 1988 Nov;51(11):1401-4. doi: 10.1136/jnnp.51.11.1401. PMID 3236018
- [Background] Lieberman MD, Eisenberger NI, Crockett MJ, Tom SM, Pfeifer JH, Way BM. Putting feelings into words: affect labeling disrupts amygdala activity in response to affective stimuli. Psychol Sci. 2007 May;18(5):421-8. doi: 10.1111/j.1467-9280.2007.01916.x. PMID 17576282
- [Background] Liu CY, Wang SJ, Fuh JL, Lin CH, Yang YY, Liu HC. The correlation of depression with functional activity in Parkinson's disease. J Neurol. 1997 Aug;244(8):493-8. doi: 10.1007/s004150050131. PMID 9309555
- [Background] Lomarev MP, Kanchana S, Bara-Jimenez W, Iyer M, Wassermann EM, Hallett M. Placebo-controlled study of rTMS for the treatment of Parkinson's disease. Mov Disord. 2006 Mar;21(3):325-31. doi: 10.1002/mds.20713. PMID 16211618
- [Background] Maeda F, Chang VY, Mazziotta J, Iacoboni M. Experience-dependent modulation of motor corticospinal excitability during action observation. Exp Brain Res. 2001 Sep;140(2):241-4. doi: 10.1007/s002210100827. PMID 11521156 (Retraction: PMID 12416532 Iacoboni M, Mazziotta J, Chang VY. Exp Brain Res. 2002 Sep;146(1):127)
- [Background] Maeda F, Keenan JP, Tormos JM, Topka H, Pascual-Leone A. Interindividual variability of the modulatory effects of repetitive transcranial magnetic stimulation on cortical excitability. Exp Brain Res. 2000 Aug;133(4):425-30. doi: 10.1007/s002210000432. PMID 10985677
- [Background] Mally J, Farkas R, Tothfalusi L, Stone TW. Long-term follow-up study with repetitive transcranial magnetic stimulation (rTMS) in Parkinson's disease. Brain Res Bull. 2004 Sep 30;64(3):259-63. doi: 10.1016/j.brainresbull.2004.07.004. PMID 15464863
- [Background] Marin RS. Apathy: a neuropsychiatric syndrome. J Neuropsychiatry Clin Neurosci. 1991 Summer;3(3):243-54. doi: 10.1176/jnp.3.3.243. PMID 1821241
- [Background] Mayeux R, Sano M, Chen J, Tatemichi T, Stern Y. Risk of dementia in first-degree relatives of patients with Alzheimer's disease and related disorders. Arch Neurol. 1991 Mar;48(3):269-73. doi: 10.1001/archneur.1991.00530150037014. PMID 2001183
- [Background] Mayeux R, Stern Y, Cote L, Williams JB. Altered serotonin metabolism in depressed patients with parkinson's disease. Neurology. 1984 May;34(5):642-6. doi: 10.1212/wnl.34.5.642. PMID 6200801
- [Background] Mayeux R, Stern Y, Williams JB, Cote L, Frantz A, Dyrenfurth I. Clinical and biochemical features of depression in Parkinson's disease. Am J Psychiatry. 1986 Jun;143(6):756-9. doi: 10.1176/ajp.143.6.756. PMID 2424323
- [Background] Mennemeier M, Triggs W, Chelette K, Woods A, Kimbrell T, Dornhoffer J. Sham Transcranial Magnetic Stimulation Using Electrical Stimulation of the Scalp. Brain Stimul. 2009 Jul 1;2(3):168-173. doi: 10.1016/j.brs.2009.02.002. PMID 20160893
- [Background] Miller KM, Okun MS, Fernandez HF, Jacobson CE 4th, Rodriguez RL, Bowers D. Depression symptoms in movement disorders: comparing Parkinson's disease, dystonia, and essential tremor. Mov Disord. 2007 Apr 15;22(5):666-72. doi: 10.1002/mds.21376. PMID 17266084
- [Background] Mir P, Matsunaga K, Gilio F, Quinn NP, Siebner HR, Rothwell JC. Dopaminergic drugs restore facilitatory premotor-motor interactions in Parkinson disease. Neurology. 2005 Jun 14;64(11):1906-12. doi: 10.1212/01.WNL.0000163772.56128.A8. PMID 15955942
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044
- [Background] Okabe S, Ugawa Y, Kanazawa I; Effectiveness of rTMS on Parkinson's Disease Study Group. 0.2-Hz repetitive transcranial magnetic stimulation has no add-on effects as compared to a realistic sham stimulation in Parkinson's disease. Mov Disord. 2003 Apr;18(4):382-8. doi: 10.1002/mds.10370. PMID 12671943
- [Background] Pascual-Leone A, Rubio B, Pallardo F, Catala MD. Rapid-rate transcranial magnetic stimulation of left dorsolateral prefrontal cortex in drug-resistant depression. Lancet. 1996 Jul 27;348(9022):233-7. doi: 10.1016/s0140-6736(96)01219-6. PMID 8684201
- [Background] Pascual-Leone A, Valls-Sole J, Brasil-Neto JP, Cammarota A, Grafman J, Hallett M. Akinesia in Parkinson's disease. II. Effects of subthreshold repetitive transcranial motor cortex stimulation. Neurology. 1994 May;44(5):892-8. doi: 10.1212/wnl.44.5.892. PMID 8190293
- [Background] Paus T, Castro-Alamancos MA, Petrides M. Cortico-cortical connectivity of the human mid-dorsolateral frontal cortex and its modulation by repetitive transcranial magnetic stimulation. Eur J Neurosci. 2001 Oct;14(8):1405-11. doi: 10.1046/j.0953-816x.2001.01757.x. PMID 11703468
- [Background] Piasecki SD, Jefferson JW. Psychiatric complications of deep brain stimulation for Parkinson's disease. J Clin Psychiatry. 2004 Jun;65(6):845-9. doi: 10.4088/jcp.v65n0617. PMID 15291663
- [Background] Rickards H. Depression in neurological disorders: Parkinson's disease, multiple sclerosis, and stroke. J Neurol Neurosurg Psychiatry. 2005 Mar;76 Suppl 1(Suppl 1):i48-52. doi: 10.1136/jnnp.2004.060426. No abstract available. PMID 15718222
- [Background] Robertson EM, Theoret H, Pascual-Leone A. Studies in cognition: the problems solved and created by transcranial magnetic stimulation. J Cogn Neurosci. 2003 Oct 1;15(7):948-60. doi: 10.1162/089892903770007344. PMID 14614806
- [Background] Sackheim HA. The cognitive effectsd of electroconvulsive therapy. Cognitive Disorders: Pathophysiology and Treatment. Moos WH and Gamzu ER. New York, Marcel Decker: 183-228, 1992.
- [Background] Sawabini KA, Watts RL. Treatment of depression in Parkinson's disease. Parkinsonism Relat Disord. 2004 May;10 Suppl 1:S37-41. doi: 10.1016/j.parkreldis.2004.02.002. PMID 15109585
- [Background] Schiffer RB, Kurlan R, Rubin A, Boer S. Evidence for atypical depression in Parkinson's disease. Am J Psychiatry. 1988 Aug;145(8):1020-2. doi: 10.1176/ajp.145.8.1020. PMID 3394854
- [Background] Siebner HR. Simultaneous repetitive transcranial magnetic stimulation does not speed fine movement in PD. Neurology. 2000 Jan 11;54(1):272; author reply 273. doi: 10.1212/wnl.54.1.272-a. No abstract available. PMID 10636177
- [Background] Siebner HR, Filipovic SR, Rowe JB, Cordivari C, Gerschlager W, Rothwell JC, Frackowiak RS, Bhatia KP. Patients with focal arm dystonia have increased sensitivity to slow-frequency repetitive TMS of the dorsal premotor cortex. Brain. 2003 Dec;126(Pt 12):2710-25. doi: 10.1093/brain/awg282. Epub 2003 Aug 22. PMID 12937071
- [Background] Siebner HR, Mentschel C, Auer C, Conrad B. Repetitive transcranial magnetic stimulation has a beneficial effect on bradykinesia in Parkinson's disease. Neuroreport. 1999 Feb 25;10(3):589-94. doi: 10.1097/00001756-199902250-00027. PMID 10208595
- [Background] Snaith RP, Baugh SJ, Clayden AD, Husain A, Sipple MA. The Clinical Anxiety Scale: an instrument derived from the Hamilton Anxiety Scale. Br J Psychiatry. 1982 Nov;141:518-23. doi: 10.1192/bjp.141.5.518. No abstract available. PMID 7150890
- [Background] Squire LR, Zouzounis JA. Self-ratings of memory dysfunction: different findings in depression and amnesia. J Clin Exp Neuropsychol. 1988 Dec;10(6):727-38. doi: 10.1080/01688638808402810. PMID 3235647
- [Background] Stallings LE, Speer AM, et al. Combining SPECT and repetitive transcranial magnetic stimulation (rTMS)-left prefrontal stimulation decreases relative perfusion locally in a dose dependent manner. Neuroimage 5: S521 Abstract, 1997.
- [Background] Starkstein SE, Mayberg HS, Preziosi TJ, Andrezejewski P, Leiguarda R, Robinson RG. Reliability, validity, and clinical correlates of apathy in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 1992 Spring;4(2):134-9. doi: 10.1176/jnp.4.2.134. PMID 1627973
- [Background] Starkstein SE, Preziosi TJ, Forrester AW, Robinson RG. Specificity of affective and autonomic symptoms of depression in Parkinson's disease. J Neurol Neurosurg Psychiatry. 1990 Oct;53(10):869-73. doi: 10.1136/jnnp.53.10.869. PMID 2266368
- [Background] Strafella AP, Paus T, Barrett J, Dagher A. Repetitive transcranial magnetic stimulation of the human prefrontal cortex induces dopamine release in the caudate nucleus. J Neurosci. 2001 Aug 1;21(15):RC157. doi: 10.1523/JNEUROSCI.21-15-j0003.2001. PMID 11459878
- [Background] Strafella AP, Paus T, Fraraccio M, Dagher A. Striatal dopamine release induced by repetitive transcranial magnetic stimulation of the human motor cortex. Brain. 2003 Dec;126(Pt 12):2609-15. doi: 10.1093/brain/awg268. Epub 2003 Aug 22. PMID 12937078
- [Background] Talairach J, Tournoux P. Co-planar Stereotaxic Atlas of the Human Brain. New York, Thieme Medical Publishers, Inc. 1988.
- [Background] Tergau F, Wanschura V, Canelo M, Wischer S, Wassermann EM, Ziemann U, Paulus W. Complete suppression of voluntary motor drive during the silent period after transcranial magnetic stimulation. Exp Brain Res. 1999 Feb;124(4):447-54. doi: 10.1007/s002210050640. PMID 10090656
- [Background] Tergau F, Wassermann EM, Paulus W, Ziemann U. Lack of clinical improvement in patients with Parkinson's disease after low and high frequency repetitive transcranial magnetic stimulation. Electroencephalogr Clin Neurophysiol Suppl. 1999;51:281-8. No abstract available. PMID 10590961
- [Background] Tormos JM, Catala MD, et al. Effects of repetitive transcranial magnetic stimulation (rTMS) on EEG. Neurology 50: A317-A318 Abstract, 1998.
- [Background] Triggs WJ, McCoy KJ, Greer R, Rossi F, Bowers D, Kortenkamp S, Nadeau SE, Heilman KM, Goodman WK. Effects of left frontal transcranial magnetic stimulation on depressed mood, cognition, and corticomotor threshold. Biol Psychiatry. 1999 Jun 1;45(11):1440-6. doi: 10.1016/s0006-3223(99)00031-1. PMID 10356626
- [Background] Valero-Cabre A, Payne BR, Rushmore J, Lomber SG, Pascual-Leone A. Impact of repetitive transcranial magnetic stimulation of the parietal cortex on metabolic brain activity: a 14C-2DG tracing study in the cat. Exp Brain Res. 2005 May;163(1):1-12. doi: 10.1007/s00221-004-2140-6. Epub 2005 Feb 2. PMID 15688174
- [Background] Veazey C, Aki SO, Cook KF, Lai EC, Kunik ME. Prevalence and treatment of depression in Parkinson's disease. J Neuropsychiatry Clin Neurosci. 2005 Summer;17(3):310-23. doi: 10.1176/jnp.17.3.310. PMID 16179652
- [Background] Wassermann EM, Wang B, Zeffiro TA, Sadato N, Pascual-Leone A, Toro C, Hallett M. Locating the motor cortex on the MRI with transcranial magnetic stimulation and PET. Neuroimage. 1996 Feb;3(1):1-9. doi: 10.1006/nimg.1996.0001. PMID 9345470
- [Background] Wu AD, Fregni F, Simon DK, Deblieck C, Pascual-Leone A. Noninvasive brain stimulation for Parkinson's disease and dystonia. Neurotherapeutics. 2008 Apr;5(2):345-61. doi: 10.1016/j.nurt.2008.02.002. PMID 18394576
- [Background] Ziemssen T, Reichmann H. Non-motor dysfunction in Parkinson's disease. Parkinsonism Relat Disord. 2007 Aug;13(6):323-32. doi: 10.1016/j.parkreldis.2006.12.014. Epub 2007 Mar 8. PMID 17349813
- [Derived] Brys M, Fox MD, Agarwal S, Biagioni M, Dacpano G, Kumar P, Pirraglia E, Chen R, Wu A, Fernandez H, Wagle Shukla A, Lou JS, Gray Z, Simon DK, Di Rocco A, Pascual-Leone A. Multifocal repetitive TMS for motor and mood symptoms of Parkinson disease: A randomized trial. Neurology. 2016 Nov 1;87(18):1907-1915. doi: 10.1212/WNL.0000000000003279. Epub 2016 Oct 5. PMID 27708129

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled from 6 clinical centers in the United States and 1 clinical center in Canada.
Pre-assignment Details: We enrolled 61 subjects into this study with a previous enrollment goal of 85. Interim analysis revealed that 61 subjects provided sufficient power for data analysis, therefore we stopped recruitment.
Groups:
- Double rTMS: High frequency rTMS stimulation of the bilateral primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC).
  Repetitive transcranial magnetic stimulation (rTMS): DLPFC Active rTMS: Each treatment will consist of 2000 stimuli (50 X 4-second trains of 40 stimuli at 10 Hz, administered every 30 seconds for 25 minutes). Stimulus intensity for the first and second trains will be 80 and 90 percent of motor evoked potential (MEP), respectively. If no adverse effects are observed following each of the first two trains, then the subsequent trains will be given at MEP threshold.
  M1 Active rTMS: Stimulation will be applied one side at a time, to the motor cortex site at 90 percent of each subject's motor threshold intensity, and at a frequency of 10 Hz with 1000 stimuli per side (25 X 8-second trains of 40 stimuli).
  Sham rTMS: Patients from all four centers randomized to receive sham treatment will undergo the same procedures used in patients receiving active rTMS.
- M1 Active rTMS + DLPFC Sham rTMS: High frequency stimulation of the primary motor cortex (M1) and sham stimulation of the dorsolateral prefrontal cortex (DLPFC).
  Repetitive transcranial magnetic stimulation (rTMS): DLPFC Active rTMS: Each treatment will consist of 2000 stimuli (50 X 4-second trains of 40 stimuli at 10 Hz, administered every 30 seconds for 25 minutes). Stimulus intensity for the first and second trains will be 80 and 90 percent of motor evoked potential (MEP), respectively. If no adverse effects are observed following each of the first two trains, then the subsequent trains will be given at MEP threshold.
  M1 Active rTMS: Stimulation will be applied one side at a time, to the motor cortex site at 90 percent of each subject's motor threshold intensity, and at a frequency of 10 Hz with 1000 stimuli per side (25 X 8-second trains of 40 stimuli).
  Sham rTMS: Patients from all four centers randomized to receive sham treatment will undergo the same procedures used in patients receiving active rTMS.
- DLPFC Active rTMS + M1 Sham rTMS: High frequency stimulation of the dorsolateral prefrontal cortex (DLPFC) and sham stimulation of the primary motor cortex (M1).
  Repetitive transcranial magnetic stimulation (rTMS): DLPFC Active rTMS: Each treatment will consist of 2000 stimuli (50 X 4-second trains of 40 stimuli at 10 Hz, administered every 30 seconds for 25 minutes). Stimulus intensity for the first and second trains will be 80 and 90 percent of motor evoked potential (MEP), respectively. If no adverse effects are observed following each of the first two trains, then the subsequent trains will be given at MEP threshold.
  M1 Active rTMS: Stimulation will be applied one side at a time, to the motor cortex site at 90 percent of each subject's motor threshold intensity, and at a frequency of 10 Hz with 1000 stimuli per side (25 X 8-second trains of 40 stimuli).
  Sham rTMS: Patients from all four centers randomized to receive sham treatment will undergo the same procedures used in patients receiving active rTMS.
- Double Sham rTMS: Sham rTMS stimulation of the bilateral primary motor cortex (M1) and left dorsolateral prefrontal cortex (DLPFC).
  Repetitive transcranial magnetic stimulation (rTMS): DLPFC Active rTMS: Each treatment will consist of 2000 stimuli (50 X 4-second trains of 40 stimuli at 10 Hz, administered every 30 seconds for 25 minutes). Stimulus intensity for the first and second trains will be 80 and 90 percent of motor evoked potential (MEP), respectively. If no adverse effects are observed following each of the first two trains, then the subsequent trains will be given at MEP threshold.
  M1 Active rTMS: Stimulation will be applied one side at a time, to the motor cortex site at 90 percent of each subject's motor threshold intensity, and at a frequency of 10 Hz with 1000 stimuli per side (25 X 8-second trains of 40 stimuli).
  Sham rTMS: Patients from all four centers randomized to receive sham treatment will undergo the same procedures used in patients receiving active rTMS.
Period: Overall Study
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Started | 20 | 14 | 12 | 15
Completed | 15 | 12 | 10 | 13
Not Completed | 5 | 2 | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS | Total
Number analyzed (Participants) | 20 | 14 | 12 | 15 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (8.0) | 62.7 (13.0) | 67.3 (12.7) | 66.2 (12.7) | 66.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 6 | 4 | 24
  Male | 11 | 9 | 6 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Motor Subscale of the Unified Parkinson's Disease Rating Scale (UPDRS Part III)
Description: To evaluate the motor symptoms in Parkinson's Disease.
  The UPDRS-III mean scores were reported for each group at each time point. The UPDRS-III Score Range is 0 - 56, where higher the score indicates greater severity of the motor symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 32.3 (8.9) | 33.1 (7.8) | 32.8 (10.7) | 28.9 (6.4)
  Week 1 Post-Treatment | 31.2 (12.5) | 27.4 (8.8) | 30.3 (14.6) | 28.2 (8.8)
  Month 1 Post-Treatment | 30.1 (9.4) | 28.1 (9.1) | 29.3 (11.4) | 28.6 (7.2)
  Month 3 Post-Treatment | 29.6 (10.3) | 33.2 (12.9) | 31.5 (11.3) | 28.6 (7.8)
  Month 6 Post-Treatment | 30.5 (11.5) | 30.6 (14.4) | 28.8 (10.1) | 29.0 (5.6)

2. Primary Outcome: Hamilton Depression Scale (HAM-D)
Description: To evaluate the depressive mood symptoms in PD.
  The HAM-D mean scores were reported for each group at each time point. The HAM-D Score Range is 0 - 56, where higher the score indicates greater severity of depressive mood symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 15.2 (6.0) | 16.7 (3.9) | 13.8 (4.6) | 14.1 (3.7)
  Week 1 Post-Treatment | 11.3 (6.2) | 11.2 (6.3) | 9.4 (5.9) | 9.3 (5.9)
  Month 1 Post-Treatment | 10.6 (6.9) | 10.1 (5.4) | 12.4 (8.1) | 8.0 (3.7)
  Month 3 Post-Treatment | 10.7 (6.9) | 10.1 (5.4) | 10.4 (7.4) | 11.1 (5.0)
  Month 6 Post-Treatment | 10.4 (7.5) | 8.6 (7.7) | 10.4 (4.5) | 10.4 (5.9)

3. Secondary Outcome: Clinical Anxiety Scale (CAS)
Description: To evaluate anxiety in Parkinson's Disease. The CAS mean scores were reported for each group at each time point. The CAS Score Range is 0 - 100, where higher the score indicates greater severity of the anxiety symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 36.3 (17.1) | 34.3 (14.1) | 33.4 (17.4) | 37.5 (16.8)
  Week 1 Post Treatment | 34.2 (16.7) | 31.0 (13.8) | 27.6 (17.4) | 32.4 (16.8)
  Month 1 Post Treatment | 31.7 (15.4) | 30.8 (12.9) | 30.8 (17.7) | 28.2 (15.3)
  Month 3 Post Treatment | 33.1 (17.4) | 27.3 (7.9) | 31.4 (16.7) | 28.5 (18.5)
  Month 6 Post Treatment | 33.4 (19.4) | 28.1 (10.9) | 24.8 (9.9) | 35.0 (15.9)

4. Secondary Outcome: Apathy Evaluation Scale (AES)
Description: To evaluate apathy in Parkinson's Disease. The AES mean scores were reported for each group at each time point. The AES Score Range is 0-42, where higher the score indicates greater severity of the apathy symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 15.6 (6.1) | 15.9 (7.1) | 18.7 (8.1) | 16.3 (5.7)
  Week 1 Post Treatment | 16.2 (5.1) | 16.9 (8.4) | 18.1 (8.8) | 15.5 (5.9)
  Month 1 Post Treatment | 17 (6.4) | 14.6 (8.1) | 19.0 (9.7) | 15.0 (5.3)
  Month 3 Post Treatment | 16.9 (7.4) | 15.1 (8.1) | 19.3 (9.3) | 16.1 (6.1)
  Month 6 Post Treatment | 17.8 (9.0) | 12.4 (8.5) | 15.8 (6.2) | 16.2 (5.2)

5. Secondary Outcome: Parkinson's Disease Questionnaire 39 (PDQ-39)
Description: To assess the quality of life (QOL) in Parkinson's Disease. The PDQ-39 mean scores were reported for each group at each time point. The PDQ-39 Score Range is 0 - 156, where higher the score indicates greater impact on quality of life.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 57.6 (25.4) | 61.5 (20.2) | 51.9 (27.5) | 55.5 (21.6)
  Week 1 Post Treatment | 51.2 (25.4) | 60.7 (19.4) | 46.8 (27.4) | 43.1 (20.1)
  Month 1 Post Treatment | 49.9 (23.6) | 56.8 (16.8) | 49.4 (28.1) | 40.9 (21.3)
  Month 3 Post Treatment | 51.7 (29.6) | 53.1 (13.8) | 49.4 (30.2) | 43.1 (21.7)
  Month 6 Post Treatment | 50.5 (25.7) | 48.3 (16.2) | 49 (20.3) | 47.5 (18.9)

6. Secondary Outcome: Montreal Cognitive Assessment (MoCA)
Description: To screen and follow cognitive function in Parkinson's Disease. The MoCA mean scores were reported for each group at each time point. The MoCA Score Range is 0 - 30, where 26-30 indicates normal cognition.
Time Frame: pre-treatment; 0,1,3, and 6 months post-treatment
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 28.2 (2.0) | 26.6 (2.5) | 27.3 (2.7) | 26.2 (4.3)
  Week 1 Post Treatment | 26.8 (3.9) | 27.1 (3.8) | 26.3 (4.2) | 27.8 (2.4)
  Month 1 Post Treatment | 28.8 (1.6) | 27.2 (3.5) | 26.8 (2.9) | 28.7 (0.9)
  Month 3 Post Treatment | 26.5 (8.0) | 25.3 (8.6) | 26.7 (3.3) | 24.9 (8.4)
  Month 6 Post Treatment | 28.0 (1.0) | 27.9 (1.7) | 26.6 (2.7) | 28.0 (2.4)

7. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Parts I, II, and IV
Description: To assess apathy, cognition, depression, activities of daily living (ADL), quality of life (QOL), and motor symptoms in Parkinson's Disease.
  The UPDRS I, II, IV total mean scores were reported for each group at each time point. The UPDRS I, II, IV scores were added together for each patient, with a total score range of 0 - 91, where higher the score indicates greater severity of the symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 25.4 (9.6) | 26.1 (8.8) | 21.5 (7.4) | 19.6 (6.6)
  Week 1 Post Treatment | 23.3 (9.8) | 23.2 (8.3) | 19.3 (7.1) | 15.5 (6.3)
  Month 1 Post Treatment | 21.8 (9.8) | 23.0 (8.8) | 19.9 (6.4) | 16.5 (6.8)
  Month 3 Post Treatment | 21.1 (12.1) | 23.2 (8.0) | 18.9 (7.9) | 16.9 (6.3)
  Month 6 Post Treatment | 23.8 (12.7) | 22.7 (7.2) | 20.2 (6.8) | 18.8 (6.6)

8. Secondary Outcome: Beck Depression Inventory (BDI-II)
Description: To assess mood symptoms in Parkinson's Disease. The BDI-II mean scores were reported for each group at each time point. The BDI-II Score Range is 0 - 63, where higher the score indicates greater severity of the mood symptoms.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment) | 23.2 (12.7) | 18.5 (8.3) | 21.7 (11.9) | 18.8 (8.1)
  Week 1 Post Treatment | 20.7 (12.0) | 16.5 (10.6) | 18.2 (13.7) | 13.7 (5.7)
  Month 1 Post Treatment | 16.4 (10.0) | 16.7 (10.1) | 20.2 (15.5) | 13.1 (5.5)
  Month 3 Post Treatment | 17.9 (11.8) | 19.1 (10.7) | 19.0 (15.3) | 14.7 (6.6)
  Month 6 Post Treatment | 20.1 (15.6) | 16.3 (10.8) | 15.7 (7.1) | 16.8 (7.4)

9. Secondary Outcome: Global Impression Scales
Description: To assess symptom severity and treatment response in Parkinson's Disease. The CGI mean scores were reported for each group at each time point. The CGI Score Range is 1 - 8, where higher the score indicates greater severity of illness or worsening of illness.
Time Frame: Pre-treatment; Post-treatment 0,1,3, and 6 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
units on a scale
  Baseline (Pre-Treatment): Severity | 4.9 (1.3) | 4.7 (1.5) | 4.3 (1.5) | 3.6 (2.1)
  Week 1 Post Treatment: Severity | 4.8 (0.8) | 4.9 (0.6) | 4.7 (0.6) | 3.9 (1.2)
  Week 1 Post Treatment: Improvement | 3.6 (0.9) | 3.5 (0.8) | 3.5 (1.0) | 3.0 (1.1)
  Month 1 Post Treatment: Severity | 4.4 (1.4) | 4.8 (0.6) | 4.4 (0.7) | 4.1 (0.7)
  Month 1 Post Treatment: Improvement | 3.5 (1.1) | 3.8 (0.8) | 3.7 (0.8) | 3.5 (1.3)
  Month 3 Post Treatment: Severity | 4.6 (0.8) | 3.8 (2.4) | 4.4 (0.7) | 4.4 (0.5)
  Month 3 Post Treatment: Improvement | 3.7 (0.6) | 3.4 (1.5) | 3.6 (1.1) | 3.6 (1.0)
  Month 6 Post Treatment: Severity | 4.2 (1.6) | 5.0 (0.8) | 4.3 (0.5) | 4.6 (0.5)
  Month 6 Post Treatment: Improvement | 3.5 (1.2) | 4.2 (0.8) | 3.7 (0.7) | 3.4 (1.2)

10. Secondary Outcome: The Number All Types of Adverse Events.
Description: To establish the safety and tolerability of rTMS in Parkinson's Disease.
Time Frame: Baseline through Month 6
Measure: Number; unit: incidents of an adverse event
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Number analyzed (Participants) | 20 | 14 | 12 | 15
incidents of an adverse event | 18 | 14 | 1 | 1

ADVERSE EVENTS:
Time Frame: Baseline through 6 months post-treatment.
Arm/Group | Double rTMS | M1 Active rTMS + DLPFC Sham rTMS | DLPFC Active rTMS + M1 Sham rTMS | Double Sham rTMS
Serious Adverse Events (participants affected / at risk) | 1/20 | 1/14 | 0/12 | 1/15
Other Adverse Events (participants affected / at risk) | 5/20 | 3/14 | 1/12 | 0/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double rTMS (N=20) | M1 Active rTMS + DLPFC Sham rTMS (N=14) | DLPFC Active rTMS + M1 Sham rTMS (N=12) | Double Sham rTMS (N=15)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Choking Episode (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Fall (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Determined to be unrelated to the study by overseeing physician.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double rTMS (N=20) | M1 Active rTMS + DLPFC Sham rTMS (N=14) | DLPFC Active rTMS + M1 Sham rTMS (N=12) | Double Sham rTMS (N=15)
Worsened Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Worsened Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Hospitlization (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Atrial Fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Neck Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4) | 0 (0) | 0 (0) — 2 incidents determined to be unrelated to the study by overseeing physician. 2 incident determined to be possibly related to the study by overseeing physician. 1 incident determined to be related to the study by overseeing physician.
Heart Burn (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Right-Sided Soreness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Fall (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Headache (Nervous system disorders) | 3 (5) | 2 (3) | 0 (0) | 0 (0) — Determined to be possibly related to the study by overseeing physician.
Left Hip Ache (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be possibly related to the study by overseeing physician.
Scalp Pain (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) — Determined to be related to the study by overseeing physician.
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) — 1 incident determined to be unrelated to the study by overseeing physician; 2 incidents in same participant determined to be related to the study by overseeing physician.
Worsening Dyskinesia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Determined to be possibly related to the study by overseeing physician.
Torn Ligament of R Lower Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Determined to be unrelated to the study by overseeing physician.

LIMITATIONS AND CAVEATS:
The study did not reach the enrollment goal of 120 patients reducing the statistical power of the study. Additionally, patients with mild and advanced disease with variable years of drug exposure were enrolled, which may obscure effects in subgroups.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No